CLINICAL TRIAL: NCT03167242
Title: A Phase 2 Interventional, Multicenter, Randomized Open Label Study to Determine the Effective and Tolerable Dose of KAF156 and Lumefantrine Solid Dispersion Formulation in Combination, Given Once Daily for 1, 2 and 3-days to Adults and Children With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Efficacy and Safety of KAF156 in Combination With LUM-SDF in Adults and Children With Uncomplicated Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CKAF156A2202; 2020-003284-25 (EudraCT Number)
Record Dates: First submitted 2017-05-19; First posted 2017-05-25 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-12

CONDITIONS: Acute Uncomplicated Plasmodium Falciparum Malaria
MeSH Terms: interventions — ganaplacide; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 day (Experimental): Participants received a single oral dose of KAF156 400 mg and LUM-SDF 960 mg
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 day (Experimental): Participants received a single oral dose of KAF156 800 mg and LUM-SDF 960 mg
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 days (Experimental): Participants received KAF156 400 mg and LUM-SDF 960 mg once daily via oral administration for 2 days
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 days (Experimental): Participants received KAF156 200 mg and LUM-SDF 480 mg once daily via oral administration for 3 days
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 days (Experimental): Participants received KAF156 400 mg and LUM-SDF 480 mg once daily via oral administration for 3 days
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 days (Experimental): Participants received KAF156 400 mg and LUM-SDF 960 mg once daily via oral administration for 3 days
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part A - Cohort 7: Coartem (Active Comparator): Participants received Coartem twice daily via oral administration for 3 days
  Interventions: Drug: Coartem
- PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 day (Experimental): Participants received a single oral dose of KAF156 200 mg and LUM-SDF 960 mg
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 day (Experimental): Participants received a single oral dose of KAF156 400 mg and LUM-SDF 960 mg
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 days (Experimental): Participants received KAF156 400 mg and LUM-SDF 960 mg once daily via oral administration for 2 days
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 days (Experimental): Participants received KAF156 400 mg and LUM-SDF 960 mg once daily via oral administration for 3 days
  Interventions: Drug: KAF156; Drug: Lumefantrine Solid Dispersion Formulation
- Part B - Cohort 4: Coartem (Active Comparator): Participants received Coartem twice daily via oral administration for 3 days
  Interventions: Drug: Coartem

INTERVENTIONS:
Drug: KAF156 — KAF156 comes in 100 mg tablets for oral administration. KAF156 was administered in combination with LUM-SDF once daily (QD) for 1, 2 or 3 days at 200 mg, 400 mg or 800 mg doses.
  Other Names: KAF
  Arms: PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 day; Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 day; Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 day; Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 days; Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 days; Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 days; Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 days; Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 day; Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 days; Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 days
Drug: Coartem — Coartem comes as 20/120 mg dispersible tablets or 80/480 mg tablets for oral administration. Coartem was administered twice daily for 3 days as active comparator.
  Arms: Part A - Cohort 7: Coartem; Part B - Cohort 4: Coartem
Drug: Lumefantrine Solid Dispersion Formulation — LUM-SDF comes in 240 mg or 480 mg sachets for oral administration. LUM-SDF was administered in combination with KAF156 once daily (QD) for 1, 2 or 3 days at 480 mg or 960 mg doses.
  Other Names: LUM-SDF and LUM
  Arms: PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 day; Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 day; Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 day; Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 days; Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 days; Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 days; Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 days; Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 day; Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 days; Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 days

SUMMARY:
This study was designed to determine the most effective and tolerable dose at the shortest dosing regimen of the investigational drug KAF156 in combination with a solid dispersion formulation of lumefantrine (LUM-SDF) in adult/adolescent and pediatric patients with uncomplicated Plasmodium falciparum malaria.

There is unmet medical need for anti-malarial treatment with new mechanism of action to reduce probability of developing resistance, and for duration shorter than 3 days of treatment and/or reduced pill burden.

DETAILED DESCRIPTION:
This was a Phase 2 multi-center and open-label study with a single cohort pharmacokinetic (PK) Run-in Part followed by 2 randomized parallel-group parts, Part A and Part B, in adults and children with confirmed and uncomplicated Plasmodium falciparum malaria. Each part (PK Run-in, Part A and Part B) had the same design structure: A screening phase of up to 24 hours where participants were evaluated for eligibility and randomized (Part A and B) into different cohorts. A treatment phase of up to 3 days where participants were treated for 1, 2 or 3 consecutive days. Finally, participants were followed up until Day 43, where the rescue medication was the local standard at the discretion of the Investigator and participants

PK Run-in part: Adult/adolescent participants (≥ 12 years old) were dosed with a single dose of 200 mg KAF156 and 960 mg LUM-SDF at Day 1. The purpose of this part was to assess potential PK interactions between the compounds when dosed together.

Part A: Adult/adolescent participants (≥ 12 years old) were randomized into one of seven cohorts in a 2:2:2:2:2:2:1 ratio: six KAF156 and LUM-SDF cohorts at starting doses of 400 mg and 480 mg once daily (QD) for 1 day respectively and a control arm (Coartem twice a day (BID) for 3 days). Upon completion of Part A, all the dosing groups were evaluated in an interim assessment to determine the effective and tolerated KAF156 and LUM-SDF dosing regimen and dosages to be used in Part B.

Part B: Children participants (2 to < 12 years old) were randomized to three KAF156 and LUM-SDF cohorts at dosages and dosing regimens selected from Part A and the control arm (Coartem) in a 2:2:2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Part A: male and female patients ≥ 12 years and with a body weight ≥ 35.0 kg. Part B: after determining the effective/tolerated doses and regimens in adolescent and adult patients, male and female patients ≥ 2 and < 12 years and with a body weight ≥ 10.0 kg will be included.
* Microscopic confirmation of P. falciparum by Giemsa-stained thick and thin films.
* P. falciparum parasitaemia of more than 1000 and less than 150 000 parasites/µL at the time of pre-screening (i.e., Study Visit 1).
* Axillary temperature ≥ 37.5 ºC or oral/tympanic/rectal temperature ≥ 38.3 ºC; or similar history of fever during the previous 24 hours (history of fever must be documented).
* Written informed consent must be obtained before any assessment is performed. If the patient is unable to read and write, then a witnessed consent according to local ethical standards is permitted. Patients < 18 years old, who are capable of providing assent, must provide assent with parental/legal guardian consent or as per local ethical guidelines.

Exclusion Criteria:

* Mixed Plasmodium infections.
* Signs and symptoms of severe malaria according to WHO (World Health Organization) 2015 criteria unless characterized by high parasitaemia only.
* Patients with concurrent febrile illnesses (e.g., typhoid fever).
* Severe vomiting, defined as more than 3 times in the 24 hours prior to inclusion in the study or severe diarrhea defined as more than 3 watery stools per day.
* Pregnant or nursing (lactating) women.
* Clinically relevant abnormalities of electrolyte balance which require correction, e.g., hypokalemia, hypocalcemia or hypomagnesemia.
* Anemia (Hemoglobin level < 8 g/dL).
* Patients with prior antimalarial therapy or antibiotics with antimalarial activity within minimum of their five (5) plasma half-lives (or within 4 weeks of screening if half-life is unknown).
* History or family history of long QT syndrome or sudden cardiac death, or any other clinical condition known to prolong the QTc (heart rate-corrected QT) interval, such as history of symptomatic cardiac arrhythmias, clinically relevant bradycardia or severe heart disease.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the patient in case of participation in the study. The investigator should make this determination in consideration of the patient's medical history and/or clinical or laboratory evidence of any of the following:
* AST/ALT > 2 x the upper limit of normal range (ULN), regardless of the level of total bilirubin
* AST/ALT > 1.5 and ≤ 2 x ULN and total bilirubin is > ULN
* Total bilirubin > 2 x ULN, regardless of the level of AST/ALT

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmaceuticals
Locations (11):
- Novartis Investigative Site, Nanoro, Burkina Faso
- Novartis Investigative Site, Lambaréné, Gabon
- Novartis Investigative Site, Ranchi, Jharkhand, India
- Kenya (2):
  - Novartis Investigative Site, Kombewa
  - Novartis Investigative Site, Siaya
- Novartis Investigative Site, Sotouba, Mali
- Novartis Investigative Site, Chokwé, Mozambique
- Novartis Investigative Site, Tak, Thailand
- Uganda (2):
  - Novartis Investigative Site, Masaka
  - Novartis Investigative Site, Tororo
- Novartis Investigative Site, Binh Phuoc Province, VNM, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

REFERENCES:
- [Derived] Sangana R, Ogutu B, Yeka A, Kusemererwa S, Tinto H, Toure AO, Kibuuka A, Lingani M, Lourenco C, Mombo-Ngoma G, Nduba V, Landry N'Guessan T, Nassa GJW, Nyantaro M, Tina LO, Anvikar A, Sinha A, Kaguthi G, Fofana B, Grobusch MP, Gaaloul ME, Marrast AC, Pathan R, Chikoto H, Csermak K, Risterucci C, Su G, Winnips C, Zhang J, Zack J. Pharmacokinetics of Ganaplacide and Lumefantrine in Adults, Adolescents, and Children with Plasmodium falciparum Malaria Treated with Ganaplacide Plus Lumefantrine Solid Dispersion Formulation: Analysis of Data from a Multinational Phase 2 Study. J Clin Pharmacol. 2025 Feb;65(2):179-189. doi: 10.1002/jcph.6138. Epub 2024 Sep 29. PMID 39344281
- [Derived] Ogutu B, Yeka A, Kusemererwa S, Thompson R, Tinto H, Toure AO, Uthaisin C, Verma A, Kibuuka A, Lingani M, Lourenco C, Mombo-Ngoma G, Nduba V, N'Guessan TL, Nassa GJW, Nyantaro M, Tina LO, Singh PK, El Gaaloul M, Marrast AC, Chikoto H, Csermak K, Demin I, Mehta D, Pathan R, Risterucci C, Su G, Winnips C, Kaguthi G, Fofana B, Grobusch MP. Ganaplacide (KAF156) plus lumefantrine solid dispersion formulation combination for uncomplicated Plasmodium falciparum malaria: an open-label, multicentre, parallel-group, randomised, controlled, phase 2 trial. Lancet Infect Dis. 2023 Sep;23(9):1051-1061. doi: 10.1016/S1473-3099(23)00209-8. Epub 2023 Jun 13. PMID 37327809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 13 sites in 10 countries.
Pre-assignment Details: Before being enrolled in the study, participants underwent a prescreening evaluation to ascertain the Plasmodium falciparum parasitemia count.
Period: Overall Study
Arm/Group | PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem
Started (All participants who were enrolled in the PK Run-in part or randomized in Parts A or B.) | 12 | 51 | 51 | 51 | 54 | 51 | 52 | 27 | 53 | 53 | 45 | 24
Full Analysis Set (FAS) (All enrolled participants, who received at least one dose of the study treatment) | 12 | 51 | 51 | 51 | 54 | 51 | 52 | 27 | 52 | 53 | 45 | 24
Pharmacokinetics (PK) Analysis Set (All enrolled participants with at least 80% compliance to study treatment who had evaluable PK parameter data and did not receive the prohibited medications which could impact PK parameters.) | 12 | 47 | 51 | 46 | 48 | 46 | 45 | 24 | 48 | 46 | 41 | 24
Per-Protocol Set (PPS) (All participants comprised in FAS who met predefined criteria related to protocol and treatment compliance.) | 12 | 50 | 48 | 48 | 47 | 44 | 43 | 25 | 48 | 46 | 40 | 22
Rich Pharmacokinetics (PK) Analysis Subset (Subset of participants within PK Run-in and Part A and comprised in PK Analysis set from whom rich PK data was collected.) | 12 | 5 | 6 | 6 | 6 | 12 | 5 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 50 | 48 | 50 | 53 | 49 | 50 | 26 | 52 | 53 | 43 | 23
Not Completed | 0 | 1 | 3 | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 2 | 1
Not completed — Patient/Guardian Decision | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1
Not completed — Reason not provided | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem | Total
Number analyzed (Participants) | 12 | 51 | 51 | 51 | 54 | 51 | 52 | 27 | 53 | 53 | 45 | 24 | 524
Age, Continuous [Mean (Standard Deviation); unit: Years] | 17.8 (10.25) | 22.3 (13.53) | 21.3 (10.69) | 21.1 (11.09) | 23.3 (14.68) | 20.3 (11.90) | 20.0 (9.49) | 20.9 (12.28) | 6.6 (2.86) | 6.2 (2.90) | 6.9 (2.60) | 5.9 (2.21) | 16.3 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 26 | 24 | 21 | 26 | 25 | 20 | 13 | 31 | 29 | 20 | 15 | 256
  Male | 6 | 25 | 27 | 30 | 28 | 26 | 32 | 14 | 22 | 24 | 25 | 9 | 268
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 7 | 7 | 7 | 9 | 7 | 7 | 4 | 1 | 1 | 0 | 0 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 44 | 44 | 43 | 45 | 44 | 45 | 23 | 52 | 52 | 45 | 24 | 473
  White | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A and Part B: Number of Participants With Polymerase Chain Reaction (PCR)-Corrected Adequate Clinical and Parasitological Response (ACPR) at Day 29
Description: PCR-corrected ACPR defined as the absence of parasitaemia was evaluated at Day 29 (i.e., 28 days post first dose) based on the short half-life of the study drugs. Microscopic species identification was confirmed and determined by PCR genotyping methods to establish malaria recrudescence/reinfection.
  A participant was considered as PCR-corrected ACPR at Day 29 if the participant did not meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure and was absence of parasitaemia on Day 29 irrespective of axillary temperature unless the presence of parasitaemia after 7 days was due to reinfection based on PCR. A presence of parasitaemia after 7 days of treatment initiation was considered as a reinfection only if the parasitaemia was clear before Day 8 and none of the parasite strain(s) detected on Day 8 or later matched with the parasite strain at baseline based on PCR.
Time Frame: 28 days post first dose
Population: All participants comprised in Per-protocol Set (PPS)
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem
Number analyzed (Participants) | 50 | 48 | 48 | 47 | 44 | 43 | 25 | 48 | 46 | 40 | 22
Participants | 46 | 45 | 47 | 47 | 44 | 42 | 25 | 37 | 42 | 38 | 21

2. Primary Outcome: PK Run-in: Area Under the Blood Concentration-time Curve Over the Last 24 Hours After Treatment Dose (AUC0-24h) of KAF156
Description: Pharmacokinetic (PK) parameters were calculated based on KAF156 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method. AUC0-24h was determined using non-compartmental methods.
Time Frame: 0, 1, 3, 6, 12, 18 and 24 hours post-dose
Population: Pharmacokinetics (PK) Analysis Set. Only participants with available PK data at the specified time point were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*μg/mL
Arm/Group | PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 Day
Number analyzed (Participants) | 11
hours*μg/mL | 5.35 (34.8)

3. Secondary Outcome: Part A and Part B: Number of Participants With Polymerase Chain Reaction (PCR)-Uncorrected Adequate Clinical and Parasitological Response (ACPR)
Description: PCR-uncorrected ACPR defined as the absence of parasitaemia was evaluated at days 15, 29 and 43 (i.e., 14, 28 and 42 days post first dose).
  A participant was considered as PCR-uncorrected ACPR at Days 15, 29 or 43 if the participant did not meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure and was absence of parasitaemia on Days 15, 29 or 43 irrespective of axillary temperature.
Time Frame: 14, 28 and 42 days post first dose
Population: All participants comprised in Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem
Number analyzed (Participants) | 51 | 51 | 51 | 54 | 51 | 52 | 27 | 52 | 53 | 45 | 24
Participants
  Day 14 post first dose | 49 | 47 | 51 | 53 | 50 | 51 | 27 | 51 | 52 | 43 | 24
  Day 28 post first dose | 46 | 40 | 48 | 51 | 45 | 47 | 26 | 34 | 41 | 36 | 15
  Day 42 post first dose | 42 | 36 | 45 | 45 | 41 | 45 | 19 | 29 | 33 | 31 | 11

4. Secondary Outcome: Part A and Part B: Number of Participants With Polymerase Chain Reaction (PCR)-Corrected Adequate Clinical and Parasitological Response (ACPR)
Description: PCR-corrected ACPR defined as the absence of parasitaemia was evaluated at days 15 and 43 (i.e., 14 and 42 days post first dose). Microscopic species identification was confirmed and determined by PCR genotyping methods to establish malaria recrudescence/reinfection.
  A participant was considered as PCR-corrected ACPR at Day 15 or Day 43 if the participant did not meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure and was absence of parasitaemia on Day 15 or Day 43 irrespective of axillary temperature unless the presence of parasitaemia after 7 days was due to reinfection based on PCR. A presence of parasitaemia after 7 days of treatment initiation was considered as a reinfection only if the parasitaemia was clear before Day 8 and none of the parasite strain(s) detected on Day 8 or later matched with the parasite strain at baseline based on PCR.
Time Frame: 14 and 42 days post first dose
Population: All participants comprised in Per-protocol Set (PPS)
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem
Number analyzed (Participants) | 50 | 48 | 48 | 47 | 44 | 43 | 25 | 48 | 46 | 40 | 22
Participants
  Day 14 post first dose | 48 | 46 | 48 | 47 | 44 | 43 | 25 | 47 | 45 | 40 | 22
  Day 42 post first dose | 45 | 44 | 46 | 46 | 43 | 41 | 24 | 36 | 37 | 37 | 20

5. Secondary Outcome: Part A and Part B: Number of Participants With Recrudescence Events
Description: Recrudescence is defined as appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at baseline. Recrudescence must be confirmed by PCR analysis.
Time Frame: 42 days post first dose
Population: All participants comprised in Full Analysis Set (FAS).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem
Number analyzed (Participants) | 51 | 51 | 51 | 54 | 51 | 52 | 27 | 52 | 53 | 45 | 24
Participants | 4 | 3 | 1 | 1 | 0 | 2 | 0 | 12 | 7 | 3 | 2

6. Secondary Outcome: Part A and Part B: Number of Participants With Reinfection Events
Description: Reinfection is defined as appearance of asexual parasites after clearance of initial infection with a genotype different from those parasites present at baseline. Reinfection must be confirmed by PCR analysis.
Time Frame: 42 days post first dose
Population: All participants comprised in Full Analysis Set (FAS).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem
Number analyzed (Participants) | 51 | 51 | 51 | 54 | 51 | 52 | 27 | 52 | 53 | 45 | 24
Participants | 3 | 7 | 4 | 7 | 8 | 2 | 8 | 11 | 10 | 9 | 10

7. Secondary Outcome: Part A and Part B: Fever Clearance Time (FCT)
Description: Fever Clearance Time (FCT) is defined as the time from the first dose until the first time the axillary body temperature decreased below and remained below 37.5°C axillary or 38.0°C oral/tympanic/rectal for at least a further 24 hours. In case a participant received rescue medication before (fever) clearance, the time to event was censored at the first use of rescue medication.
Time Frame: 42 days post first dose
Population: Full Analysis Set (FAS). Only participants with fever at baseline and post-baseline assessment of fever clearance at the time point were included in the analysis.
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem
Number analyzed (Participants) | 16 | 7 | 8 | 15 | 13 | 9 | 5 | 9 | 11 | 10 | 5
Hours | 18.7 (3.09) | 22.5 (6.09) | 20.3 (4.92) | 16.6 (3.48) | 17.5 (2.65) | 19.2 (2.92) | 26.3 (7.67) | 23.5 (10.26) | 17.3 (7.4) | 13.8 (3.68) | 22.9 (12.78)

8. Secondary Outcome: PK Run-in, Part A and Part B: Parasite Clearance Time (PCT)
Description: Parasite Clearance Time (PCT) is defined as the time from the first dose until the first total and continued disappearance of asexual parasite forms which remained at least a further 48 hours. In case a participant received rescue medication before (parasite) clearance, the time to event was censored at the first use of rescue medication.
Time Frame: 42 days post first dose
Population: All participants comprised in Full Analysis Set (FAS).
Measure: Mean (Standard Error); unit: Hours
Arm/Group | PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem
Number analyzed (Participants) | 12 | 51 | 51 | 51 | 54 | 51 | 52 | 27 | 52 | 53 | 45 | 24
Hours | 49.9 (4.35) | 48.4 (3.5) | 46.6 (3.93) | 39.9 (2.46) | 51.4 (3.97) | 49.7 (3.72) | 48.1 (4.24) | 50.0 (12.82) | 42.6 (2.62) | 47.0 (2.79) | 41.9 (2.58) | 35.6 (2.82)

9. Secondary Outcome: PK Run-in, Part A and Part B: Number of Participants With Parasitaemia
Description: Parasitaemia is the quantitative content of parasites in the blood determined by microscopy examination validated methods. Only Plasmodium Falciparum asexual form is used for parasitaemia assessments.
Time Frame: 12, 24 and 48 hours post last dose
Population: Full Analysis Set (FAS). Only participants with assessment of parasitaemia at the timepoint were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A - Cohort 7: Coartem | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 4: Coartem
Number analyzed (Participants) | 12 | 51 | 51 | 51 | 54 | 51 | 52 | 27 | 52 | 53 | 45 | 24
Participants
  12 hours post last dose: number analyzed (Participants) | 12 | 50 | 50 | 49 | 52 | 50 | 51 | 27 | 51 | 53 | 45 | 24
  12 hours post last dose | 12 | 46 | 46 | 44 | 52 | 49 | 49 | 22 | 48 | 48 | 42 | 22
  24 hours post last dose: number analyzed (Participants) | 12 | 49 | 51 | 51 | 54 | 50 | 50 | 27 | 51 | 52 | 44 | 24
  24 hours post last dose | 11 | 39 | 41 | 38 | 46 | 42 | 34 | 14 | 41 | 42 | 36 | 17
  48 hours post last dose: number analyzed (Participants) | 12 | 50 | 51 | 51 | 53 | 49 | 52 | 26 | 51 | 52 | 44 | 24
  48 hours post last dose | 3 | 13 | 9 | 8 | 12 | 10 | 11 | 4 | 4 | 10 | 5 | 1

10. Secondary Outcome: Part A and Part B: Area Under the Blood Concentration-time Curve Over the Last 24 Hours After Last Treatment Dose (AUC0-24h) of KAF156
Description: as for outcome 2
Time Frame: 3, 6, 18 and 24 hours post last dose
Population: Pharmacokinetics (PK) Analysis Set. Only participants with available PK data at the specified time point were included in the analysis. As per study design, AUC0-24h was not determined for Part B cohorts 2 and 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*μg/mL
Arm/Group | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days
Number analyzed (Participants) | 38 | 44 | 41 | 43 | 36 | 41 | 48 | 0 | 0
hours*μg/mL | 9.84 (41.5) | 21.7 (41.7) | 9.95 (131.9) | 5.91 (29.2) | 11 (79.3) | 10.9 (57.4) | 11 (47.7) |  |

11. Secondary Outcome: Part A and Part B: Maximum Peak Observed Concentration (Cmax) of KAF156
Description: Pharmacokinetic (PK) parameters were calculated based on KAF156 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method. Cmax was determined using non-compartmental methods.
Time Frame: 3, 6, 18, 24, 27, 30, 48, 51, 54, 68, 72 and 168 hours post last dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days | Part B - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part B - Cohort 2: KAF 400 mg and LUM 960 mg QD for 2 Days | Part B - Cohort 3: KAF 400 mg and LUM 960 mg QD for 3 Days
Number analyzed (Participants) | 39 | 44 | 40 | 43 | 36 | 41 | 48 | 46 | 41
ng/mL | 653 (43.9) | 1470 (46.5) | 1060 (83.9) | 665 (30.3) | 1470 (30.9) | 1320 (32.7) | 714 (49.4) | 1060 (48.4) | 1380 (29.7)

12. Secondary Outcome: PK Run-in and Part A: Elimination Half-life (T½) of KAF156
Description: Pharmacokinetic (PK) parameters were calculated based on KAF156 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method. T½ was determined using non-compartmental methods.
Time Frame: 0, 1, 3, 6, 12, 18, 24, 27, 30, 36, 48, 72, 96 and 168 hours post last dose
Population: Rich Pharmacokinetics (PK) Analysis subset. Only participants with available PK data at the specified time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 3: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A - Cohort 4: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 5: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A - Cohort 6: KAF 400 mg and LUM 960 mg QD for 3 Days
Number analyzed (Participants) | 11 | 4 | 6 | 4 | 2 | 9 | 2
Hours | 25.0 (8.81) | 25.4 (5.32) | 29.9 (9.95) | 31.0 (3.86) | 35.8 (19.4) | 28.4 (3.49) | 26.6 (4.15)

13. Secondary Outcome: PK Run-in and Part A (Cohorts 1 and 2): Time to Reach Maximum Blood Concentrations (Tmax) of KAF156
Description: Pharmacokinetic (PK) parameters were calculated based on KAF156 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method. Tmax was determined using non-compartmental methods.
Time Frame: 0, 1, 3, 6, 12, 18, 24, 30, 48, 96 and 168 hours post last dose
Population: Rich Pharmacokinetics (PK) Analysis subset. Only participants with available PK data at the specified time point were included in the analysis. As per study design, Tmax was only determined per PK Run-in and Part A cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PK Run-in Cohort: KAF 200 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 1: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A - Cohort 2: KAF 800 mg and LUM 960 mg QD for 1 Day
Number analyzed (Participants) | 12 | 5 | 6
Hours | 4.23 (1.55) | 39.8 (77.3) | 5.99 (3.11)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from Day 1 to Day 43, where Day 43 could be 42, 41 or 40 days after end of treatment depending on whether the participant received treatment during 1, 2 or 3 consecutive days respectively.
Description: Any sign or symptom that occurs during the study treatment plus the 40, 41 or 42 days post treatment depending on whether the participant received treatment during 1, 2 or 3 consecutive days respectively.
  Part A and Part B safety data was pooled for safety analysis since Part B cohorts 1, 2 and 3 dosages and dosing regimens match with Part A cohorts 1, 3 and 6 respectively. Part B dosages and dosing regimens were selected based on the outcome of the interim assessment in Part A.
Groups:
- PK Run-in: KAF 200 mg and LUM 960 mg QD for 1 Day: PK Run-in participants received a single oral dose of KAF156 200 mg and LUM-SDF 960 mg
- Part A: KAF 800 mg and LUM 960 mg QD for 1 Day: Part A - Cohort 2 participants received a single oral dose of KAF156 800 mg and LUM-SDF 960 mg
- Part A: KAF 200 mg and LUM 480 mg QD for 3 Days: Part A - Cohort 4 participants received KAF156 200 mg and LUM-SDF 480 mg once daily via oral administration for 3 days
- Part A: KAF 400 mg and LUM 480 mg QD for 3 Days: Part A - Cohort 5 participants received KAF156 400 mg and LUM-SDF 480 mg once daily via oral administration for 3 days
- Part A and Part B: KAF 400 mg and LUM 960 mg QD for 1 Day: Part A - Cohort 1 and Part B - Cohort 1 participants received a single oral dose of KAF156 400 mg and LUM-SDF 960 mg
- Part A and Part B: KAF 400 mg and LUM 960 mg QD for 2 Days: Part A - Cohort 3 and Part B - Cohort 2 participants received KAF156 400 mg and LUM-SDF 960 mg once daily via oral administration for 2 days
- Part A and Part B: KAF 400 mg and LUM 960 mg QD for 3 Days: Part A - Cohort 6 and Part B - Cohort 3 participants received KAF156 400 mg and LUM-SDF 960 mg once daily via oral administration for 3 days
- Part A and Part B: Coartem: Part A - Cohort 7 and Part B - Cohort 4 participants received Coartem twice daily via oral administration for 3 days
Arm/Group | PK Run-in: KAF 200 mg and LUM 960 mg QD for 1 Day | Part A: KAF 800 mg and LUM 960 mg QD for 1 Day | Part A: KAF 200 mg and LUM 480 mg QD for 3 Days | Part A: KAF 400 mg and LUM 480 mg QD for 3 Days | Part A and Part B: KAF 400 mg and LUM 960 mg QD for 1 Day | Part A and Part B: KAF 400 mg and LUM 960 mg QD for 2 Days | Part A and Part B: KAF 400 mg and LUM 960 mg QD for 3 Days | Part A and Part B: Coartem
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/51 | 0/54 | 0/51 | 0/103 | 0/104 | 0/97 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/51 | 2/54 | 1/51 | 7/103 | 5/104 | 2/97 | 3/51
Other Adverse Events (participants affected / at risk) | 7/12 | 37/51 | 30/54 | 32/51 | 69/103 | 68/104 | 59/97 | 30/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PK Run-in: KAF 200 mg and LUM 960 mg QD for 1 Day (N=12) | Part A: KAF 800 mg and LUM 960 mg QD for 1 Day (N=51) | Part A: KAF 200 mg and LUM 480 mg QD for 3 Days (N=54) | Part A: KAF 400 mg and LUM 480 mg QD for 3 Days (N=51) | Part A and Part B: KAF 400 mg and LUM 960 mg QD for 1 Day (N=103) | Part A and Part B: KAF 400 mg and LUM 960 mg QD for 2 Days (N=104) | Part A and Part B: KAF 400 mg and LUM 960 mg QD for 3 Days (N=97) | Part A and Part B: Coartem (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PK Run-in: KAF 200 mg and LUM 960 mg QD for 1 Day (N=12) | Part A: KAF 800 mg and LUM 960 mg QD for 1 Day (N=51) | Part A: KAF 200 mg and LUM 480 mg QD for 3 Days (N=54) | Part A: KAF 400 mg and LUM 480 mg QD for 3 Days (N=51) | Part A and Part B: KAF 400 mg and LUM 960 mg QD for 1 Day (N=103) | Part A and Part B: KAF 400 mg and LUM 960 mg QD for 2 Days (N=104) | Part A and Part B: KAF 400 mg and LUM 960 mg QD for 3 Days (N=97) | Part A and Part B: Coartem (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 5 | 3 | 5 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 2 | 0 | 1 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 5 | 1 | 1 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 4 | 1 | 0 | 4 | 1 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 2 | 7 | 3 | 5 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 1 | 2 | 1 | 3 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 8 | 2 | 3 | 8 | 9 | 8 | 2
Pyrexia (General disorders) | 0 | 5 | 4 | 6 | 20 | 18 | 9 | 13
Treatment failure (General disorders) | 0 | 3 | 3 | 2 | 3 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 3 | 2 | 0
Infection parasitic (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Malaria (Infections and infestations) | 0 | 8 | 4 | 6 | 28 | 25 | 16 | 18
Upper respiratory tract infection (Infections and infestations) | 0 | 6 | 5 | 3 | 15 | 12 | 12 | 5
Blood phosphorus increased (Investigations) | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 5 | 9 | 9 | 5 | 6 | 9 | 3
Headache (Nervous system disorders) | 0 | 10 | 15 | 7 | 16 | 13 | 14 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 5 | 7 | 10 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT03167242/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT03167242/SAP_001.pdf